CLINICAL TRIAL: NCT05763342
Title: An Early Feasibility, Prospective, Exploratory Study Investigating the Use of Objective Measures to Inform Focused Multipolar Fitting in Adult Cochlear Implant Recipients
Brief Title: A Study of Objective Fitting for Focused Multipolar Stimulation
Acronym: OFIT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cochlear (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: AI5817
Record Dates: First submitted 2023-01-31; First posted 2023-03-10 (Actual); Last update posted 2026-02-09 (Actual); Status verified 2026-02

CONDITIONS: Hearing Loss, Bilateral
MeSH Terms: conditions — Hearing Loss, Bilateral

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Adult Cochlear Implant (Experimental): Adult cochlear implant recipients receiving different focused multipolar maps that are programmed using either behavioural or objective methods
  Interventions: Device: The Phoenix Research System

INTERVENTIONS:
Device: The Phoenix Research System — Focused Multipolar Stimulation (FMS) strategy in adult cochlear implant recipients.

SUMMARY:
The purpose of this exploratory study is to trial various objective and behavioural fitting methods for potential use with Focused Multipolar Stimulation programming.

DETAILED DESCRIPTION:
This study will compare various objective and behavioural fitting methods for the programming of Focused Multipolar Stimulation. Fitting methods will be assessed for both performance and clinician-rated experience to determine the most practical and beneficial method to balance ease of fitting and performance. Focused Multipolar Stimulation (FMS) is an alternative to the standard of care Monopolar Stimulation (MP). FMS may improve spectral resolution through reduced cochlear spread of excitation and in turn provide enhanced speech perception and real-world clinical improvement over MP stimulation.

ELIGIBILITY:
Inclusion Criteria:

1. Moderately severe to profound sensorineural hearing loss in both ears. (i.e., >55 dB HL pure-tone average loss)
2. Candidate for unilateral cochlear implantation according to locally approved criteria.
3. Aged 18 years or over.
4. Fluent speaker in the language used to assess speech perception performance.
5. Willing and able to provide written informed consent.

Exclusion Criteria:

1. Unable or unwilling to comply with the requirements of the clinical investigation as determined by the Investigator.
2. Investigator site personnel directly affiliated with this study and/or their immediate families; immediate family is defined as a spouse, parent, child, or sibling.
3. Cochlear employees or employees of Contract Research Organisations or contractors engaged by Cochlear for the purposes of this investigation.
4. Pregnant at the time of surgery.
5. Prisoners, or anyone in custody.
6. Current participation, or participation in another interventional clinical study/trial in the past 30 days, involving an investigational drug or device.
7. Previous or existing cochlear-implant recipient.
8. Evidence of severe or greater sensorineural hearing loss in the ear to be implanted prior to five years of age.
9. Duration of severe to profound hearing loss >20 years in the ear to be implanted.
10. Ossification or other cochlear anomaly that might prevent complete insertion of the electrode array.
11. Diagnosis of auditory neuropathy.
12. Deafness due to lesions of the acoustic nerve or central auditory pathway.
13. Additional handicaps that would prevent or restrict participation in the audiological evaluations.
14. Unrealistic expectations on the part of the subject regarding the possible benefits, risks, and limitations that are inherent to the surgical procedure and prosthetic device.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2024-02-08 (Actual); Primary Completion 2025-10-20 (Actual); Study Completion 2025-11-26 (Actual)

PRIMARY OUTCOMES:
Speech reception threshold (SRT) in noise as a signal-to-noise ratio for 50% correct score. | 6 months
  Difference in speech reception threshold (SRT) between objectively fit and behaviourally fit maps using the Spanish Hearing in Noise Test (HINT) to measure the SRT, reported as a signal-to-noise ratio for 50% correct score.

CONTACTS AND LOCATIONS:
Locations (1):
- Complejo Hospitalario Universitario Insular Materno Infantil de Gran Canaria, Las Palmas de Gran Canaria, Las Palmas, Spain